CLINICAL TRIAL: NCT04665713
Title: Effect of Prevalence of Overweight and Obesity(Body Mass Index (BMI)) on Efficacy of Herbal Medicines(ZiYinXieHuo) in Girls' Sexual Precocity
Brief Title: Effect of Prevalence of BMI on Efficacy of Herbal Medicines in Girls' Sexual Precocity
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ZY3-RCPY-2-2021
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Precocious Puberty
Keywords: Puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: children whose BMI are in the normal range(From P5 to P85)
- Overweight: children whose BMI are above the normal range(over P85)

SUMMARY:
Effect of Prevalence of Overweight and Obesity(Body Mass Index (BMI)) on Efficacy of herbal medicines(ZiYinXieHuo) in girls sexual Precocity

DETAILED DESCRIPTION:
Herbal medicines(ZiYinXieHuo) might have implications for the effects of treatment. in sexual Precocity among the higher BMI girls. Thus the investigator use cohort studies to confirm this hypothesis. Selected children were from the precocious puberty clinic of the affiliated Pediatrics Hospital of Fudan University. Calculated according to the sample size (sample 6), the total number of cases was 192. All cases met the selected criteria. The subjects were divided into three groups according to the cut-off point of BMI of height and weight of Chinese children and adolescents (girls age in 2-18). Compared with children of the same age and sex, overweight group includes those BMI in the range of P85-P95, obese group includes those BMI greater than (or equal to) P95, and the girls whose BMI in the range of P5-P85 are assigned to the normal group. Chinese herbs for ZiYinXieHuo were used to treat girls with precocious puberty, only given by hospital preparation, drug dose: 30ml/once, 3 times a day. A course of treatment lasts for three months. In this study, two courses of treatment (6 months） were observed. The subjects would received three examinations: before taking the drug (baseline), the third month (metaphase) and the sixth month (end point).

ELIGIBILITY:
Inclusion Criteria:

- no abnormal weight and height in parents and families, no organic diseases, no drugs affecting gonadal axis or obesity; normal health, no secondary obesity caused by endocrine and genetic metabolic diseases, no lifestyle intervention to treat obesity.

Exclusion Criteria:

- central neoplastic lesions, rare syndrome, severe heart, liver and kidney diseases and other chronic diseases such as tuberculosis, asthma, rheumatism, complicated infection, congenital hypothyroidism associated with precocious puberty, peripheral precocious puberty, incomplete precocious puberty and so on.

Ages: 4 Years to 8 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Precocious puberty is more common in girls than boys
Study Population: Selected children were from the precocious puberty clinic of the affiliated Pediatrics Hospital of Fudan University.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Bone Age | From enrollment to the sixth month after treatment
  growth of the difference between bone age and actual age after 6 months of treatment (in years)

SECONDARY OUTCOMES:
Ovarian Volume | From enrollment to the sixth month after treatment
  development of uterine volume and ovarian volume after 6 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Subspecialty Group of Endocrinologic, Hereditary and Metabolic Diseases, the Society of Pediatrics, Chinese Medical Association; Editorial Board, Chinese Journal of Pediatrics. [Consensus statement For the diagnosis and treatment of central precocious puberty (2015)]. Zhonghua Er Ke Za Zhi. 2015 Jun;53(6):412-8. No abstract available. Chinese. PMID 26310550
- [Background] Marshall WA, Tanner JM. Variations in pattern of pubertal changes in girls. Arch Dis Child. 1969 Jun;44(235):291-303. doi: 10.1136/adc.44.235.291. No abstract available. PMID 5785179
- [Background] Fugl L, Hagen CP, Mieritz MG, Tinggaard J, Fallentin E, Main KM, Juul A. Glandular breast tissue volume by magnetic resonance imaging in 100 healthy peripubertal girls: evaluation of clinical Tanner staging. Pediatr Res. 2016 Oct;80(4):526-30. doi: 10.1038/pr.2016.125. Epub 2016 Jun 3. PMID 27384405
- [Background] Sheth SS, Hajari AR, Lulla CP, Kshirsagar D. Sonographic evaluation of uterine volume and its clinical importance. J Obstet Gynaecol Res. 2017 Jan;43(1):185-189. doi: 10.1111/jog.13189. Epub 2016 Dec 8. PMID 27928854
- [Result] Group of China Obesity Task Force. [Body mass index reference norm for screening overweight and obesity in Chinese children and adolescents]. Zhonghua Liu Xing Bing Xue Za Zhi. 2004 Feb;25(2):97-102. Chinese. PMID 15132858
- [Result] Li H, Ji CY, Zong XN, Zhang YQ. [Body mass index growth curves for Chinese children and adolescents aged 0 to 18 years]. Zhonghua Er Ke Za Zhi. 2009 Jul;47(7):493-8. Chinese. PMID 19951508
- [Result] Li H, Zong XN, Ji CY, Mi J. [Body mass index cut-offs for overweight and obesity in Chinese children and adolescents aged 2 - 18 years]. Zhonghua Liu Xing Bing Xue Za Zhi. 2010 Jun;31(6):616-20. Chinese. PMID 21163089